CLINICAL TRIAL: NCT04243356
Title: Impact of Intensive Care Unit Nurse Participation in Post - ICU (Intensive Care Unit) Follow Up Clinic
Brief Title: Impact of Intensive Care Unit Nurse Participation in Post - ICU Follow Up Clinic
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jakob McSparron, Clinical Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00170939
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Nurse-Patient Relations; Nurse Role

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Encounter Group (Experimental): Nurses that are assigned to this group will be asked to take surveys before and immediately following the post-ICU clinic encounter with a patient that they had cared for in the ICU during a follow-up care visit with the former ICU - patient.
  Interventions: Behavioral: Nurse Encounter Group
- Nurse Control Group (Other): Nurses assigned to this group will only complete surveys and will not see a former patient in a post-ICU visit.
  Interventions: Other: Nurse control group

INTERVENTIONS:
Behavioral: Nurse Encounter Group — Nurses in this group will meet with former ICU patients in a post ICU clinic visit. This will be a structured meeting for approximately 15 minutes with the nurse and former patient. The encounter will be observed by a member of the research team. Surveys will be completed before and after the visits. Additionally, nurses will be interviewed 4-7 days after meeting with their former patients.
  Arms: Nurse Encounter Group
Other: Nurse control group — This group will complete surveys.
  Arms: Nurse Control Group

SUMMARY:
The objective of this study is to learn more about the impact of a longitudinal encounter between critical care nurses and former intensive care unit patients. This study will enroll 10 patients that had been admitted in an ICU to meet with a former nurse that had taken care of them in the ICU. The study will enroll 20 nurses that had taken care of these patients in the ICU. The study will randomize 10 nurses to be in the encounter group and 10 nurses to be assigned to the control group. Only nurses assigned to the encounter group will meet with the patients at their post-ICU clinic.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Patients that were admitted to the ICU that are appropriate for follow-up.

Nurses:

Inclusion Criteria:

* Registered nurse in an intensive care unit and took care of the enrolled patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in medical ICU nurse fulfillment toward the ICU following an encounter with a former ICU patient in the post-ICU clinic using an adapted Stanford Professional Fulfillment Index | Baseline, at the follow-up ICU clinic visit for the encounter group (approximately 2-4 weeks after discharge)
  The survey consists of 6 questions that are measured on a 5 point Likert scale (scored 0 to 4, with 4 representing higher fulfillment). The scores for all 6 fulfillment questions are then averaged for a composite score for fulfillment (also ranging from 0-4). The surveys will be administered at the time of enrollment for both the encounter and control nurse groups. The post-intervention survey will be administered only to the encounter group immediately following the post-ICU clinic encounter.

SECONDARY OUTCOMES:
Change in medical ICU nurse burnout following an encounter with a former ICU patient in the post-ICU clinic | Baseline, at the follow-up ICU clinic visit for the encounter group (approximately 2-4 weeks after discharge)
  The survey includes 2 questions and is adapted from Maslach Burnout Inventory (MBI) and are single-item measures of emotional exhaustion and depersonalization.
  The assessment of burnout are measured on a 7 point Likert scale (scored 0 to 6, with 6 representing higher burnout). The surveys will be administered at the time of enrollment for both the encounter and control nurse groups. The post-intervention survey will be administered only to the encounter group immediately following the post-ICU clinic encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob McSparron, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No